CLINICAL TRIAL: NCT05506189
Title: A Prospective Study on the Effect of Quality of Life and Life Style Modification for Breast Cancer Survivors Using Mobile App-based Human Coaching Program
Brief Title: Life Style Modification for Breast Canccer Survivors Using Mobile App-based Human Coaching Program
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, So-Youn Jung, Breast Surgeon, National Cancer Center, Korea
Other Study IDs: NCC 2019-0098
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer Survivors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer survivors with over-weight or obesity: Breast cancer survivors with 25 and more than 25 of BMI will be supported with 6 months life style modification program using mobile application including human coach for reducing BMI.
  Interventions: Other: mobile application program with human coach

INTERVENTIONS:
Other: mobile application program with human coach — 6-months mobile application program with human coach for life-style modifiation including diet and exercise

SUMMARY:
This study is aimed to investigate whether mobile app-based human coaching program for 6 months is effective for reducing BMI in breast cancer survivors with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

1. breast cancer survivors who have completed acute treatment of breast cancer
2. Age: 18 ~ 70 year old
3. stage: I, II, III
4. BMI≥25.0 Kg/m2
5. breast cancer survovrs who can use mobile application program
6. breast cancer survovrs who agree with this study's consent

Exclusion Criteria:

1. Stage IV, carcinoma in situ
2. breast cancer survivors who don't use smartphone
3. breast cancer survivors with previous other malignant disease
4. breast cancer survivors with multiple malignancies
5. breast cancer survivors with uncontrolled chronic comorbid disease
6. breast cancer survovrs who disagree with this study's consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer survivors with 25 and more than 25 of BMI
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
reduction of body mass index (BMI) | Baseline and 6 month
  whether the 6-month mobile program can be effective for reducing BMI

CONTACTS AND LOCATIONS:
Overall Officials: So-Youn Jung, MD PhD, Principal Investigator — Center for Breast Cancer, National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea